CLINICAL TRIAL: NCT07129252
Title: A Phase 1/2 Dose Escalation Study of CRN09682 With an Expansion Phase in Participants With Progressive Metastatic Somatostatin Receptor Type 2 (SST2)-Expressing Neuroendocrine Neoplasms (NENs) and Other SST2-Expressing Solid Tumors
Brief Title: A Study to Investigate Safety and Effectiveness of CRN09682 in Participants With SST2-Expressing NENs and Other Solid Tumors
Acronym: BRAVESST2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRN09682-191
Record Dates: First submitted 2025-07-01; First posted 2025-08-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: SST2-positive Neuroendocrine Neoplasms; Neuroendocrine Tumors; Neuroendocrine Neoplasm
Keywords: CRN09682; Crinetics; Neuroendocrine Neoplasm; NEN; Neuroendocrine Tumor; NET; MMAE; SST2; Somatostatin; Metastatic; Solid Tumor; Dose Escalation; Dose Expansion; Phase 1; SSTR+; Phase 2; Phase 1/2; Neuroendocrine Carcinoma; NEC
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasm Metastasis; Carcinoma, Neuroendocrine

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2, 2-part, multicenter, open-label, nonrandomized, multiple-dose, first-in-human study (with dose escalation and expansion phase) of CRN09682 in participants with NENs and other solid tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Experimental): Multiple Dose Levels administered Q3W
  Interventions: Drug: CRN09682
- Dose Expansion: Cohort 1 (Experimental): Pancreatic Neuroendocrine Tumor (NET)
  Interventions: Drug: CRN09682
- Dose Expansion: Cohort 2 (Experimental): Non-Pancreatic NET
  Interventions: Drug: CRN09682
- Dose Expansion: Cohort 3 (Experimental): Neuroendocrine Carcinoma (NEC)
  Interventions: Drug: CRN09682
- Dose Expansion: Cohort 4 (Experimental): Other Solid Tumors
  Interventions: Drug: CRN09682

INTERVENTIONS:
Drug: CRN09682 — Study drug CRN09682 intravenously

SUMMARY:
This Phase 1/2, multicenter, open-label, FIH study aims to evaluate the safety, tolerability, PK, and preliminary antitumor activity of CRN09682 in participants with SST2-expressing NENs and other solid tumors. The study includes a Dose Escalation Phase to determine the MTD and DLTs. Following MTD identification, additional participants will be enrolled at the expansion dose to further assess safety, tolerability, PK, and antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Have a histological diagnosis of metastatic or locally advanced inoperable NET, NEC, or other solid tumors that have confirmed radiological progression.
* Have one or more measurable disease location per RECIST version 1.1.
* Have a tumor that expresses SSR confirmed by SSR imaging.
* Have an ECOG performance status of 0, 1, or 2.

Exclusion Criteria:

* Have tumor progression while undergoing a course of PRRT or within 6 months of completing PRRT.
* Have brain metastases unless asymptomatic and stable for at least one month for participants with SCLC or LCLC or at least 3 months for participants with other non-NET solid tumors.
* Use of anticancer agents within specified intervals prior to the first dose of study drug.
* Had surgery, chemoembolization, or radiofrequency ablation within 90 days prior to first dose of study drug.
* Prior participation in any intervention clinical study within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
* Participants with carcinoid syndrome.
* Secondary malignancy: participants who have any other malignancy known to be active or treated within 3 years of the start of screening, with the exception of treated cervical intraepithelial neoplasia, superficial (noninvasive) bladder cancer, and non-melanoma skin cancer.
* Have prior treatment with MMAE.
* Have hypersensitivity or history of anaphylactic reaction to octreotide, other SSAs, and/or MMAE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
(Dose Escalation) Incidence and severity of DLTs. | From first dose through Day 21.
(Dose Escalation) Incidence and severity of AEs and SAEs at each dose level and incidence of AEs leading to discontinuation from study drug. | From first dose of study drug to 30 days after the last dose.
(Dose Expansion) Nature, incidence, and severity of AEs and SAEs at the Expansion Dose. | From first dose of study drug to 30 days after the last dose.
(Dose Expansion) Interruptions at the Expansion Dose. | At Day 1 of each cycle through study completion, approximately 2 years.

SECONDARY OUTCOMES:
(Dose Escalation) Maximum Plasma Concentration (Cmax) of CRN09682 and MMAE . | Day 1 of each cycle (each cycle is 21 days) for the duration of the study, from baseline to safety follow-up visit, up to 2 years.
(Dose Escalation) Time to Maximum Concentration (Tmax) of CRN09682 and MMAE. | Day 1 of each cycle (each cycle is 21 days) for the duration of the study, from baseline to safety follow-up visit, up to 2 years.
(Dose Escalation) Measure of CRN09682 and MMAE exposure in the body from initial dose to the last measurable concentration (AUC0-last). | Day 1 of each cycle (each cycle is 21 days) for the duration of the study, from baseline to safety follow-up visit, up to 2 years.
(Dose Escalation) Measure of total CRN09682 exposure in the body across time (AUC0-inf). | Day 1 of each cycle (each cycle is 21 days) for the duration of the study, from baseline to safety follow-up visit, up to 2 years.
(Dose Escalation) The amount of time required for CRN09682 to be reduced to half of its initial concentration in the blood (t1/2). | Day 1 of each cycle (each cycle is 21 days) for the duration of the study, from baseline to safety follow-up visit, up to 2 years.
(Dose Escalation & Expansion) Objective response rate (ORR): The percentage of patients with best overall response of complete response or partial response according to RECIST 1.1 | Throughout the study until disease progression or the last evaluable assessment in the absence of progression whichever occurs first, approximately 2 years.
(Dose Escalation & Expansion) Disease control rate (DCR): The percentage of patients with best overall response of complete response, partial response, or stable disease according to RECIST 1.1 | Throughout the study until disease progression or the last evaluable assessment in the absence of progression whichever occurs first , approximately 2 years.
(Dose Escalation & Expansion) Duration of response (DOR): The time from the date of first objective response until date of disease progression or death in the absence of disease progression, according to RECIST 1.1. | From the first documented objective response to disease progression or death whichever occurs first, approximately 2 years.
(Dose Expansion) Changes in somatostatin receptor imaging: Evaluate changes in SSR tracer uptake over time, based on whether uptake is greater than or less than liver uptake. | Throughout the study at predefined intervals, approximately 2 years.
(Dose Expansion) Radiographic PFS: The time from the start of study drug until RECIST 1.1 defined disease progression or death in the absence of disease progression. | Throughout the study until disease progression or death whichever occurs first, approximately 2 years.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (15):
  - Crinetics Study Site, Duarte, California
  - Crinetics Study Site, Newport Beach, California
  - Crinetics Study Site, Denver, Colorado
  - Crinetics Study Site, New Haven, Connecticut
  - Crinetics Study Site, Atlanta, Georgia
  - Crinetics Study Site, Lexington, Kentucky
  - Crinetics Study Site, Metairie, Louisiana
  - Crinetics Study Site, Grand Rapids, Michigan
  - Crinetics Study Site, Philadelphia, Pennsylvania
  - Crinetics Study Site, Austin, Texas
  - Crinetics Study Site, Houston, Texas
  - Crinetics Study Site, Irving, Texas
  - Crinetics Study Site, Salt Lake City, Utah
  - Crinetics Study Site, Charlottesville, Virginia
  - Crinetics Study Site, Fairfax, Virginia
- Spain (2):
  - Crinetics Study Site, Barcelona
  - Crinetics Study Site, Madrid

IPD SHARING:
Plan to Share IPD: No